CLINICAL TRIAL: NCT01778062
Title: A Phase Ⅲb, Multicenter, Double-blind, Randomized, Controlled Trial, to Assess the Efficacy and Safety of Indacaterol (150㎍ o.d.) vs. Placebo, in Patients With Moderate-to-severe COPD With Destroyed Lung by Tuberculosis
Brief Title: Indacaterol EfectIveness In COPD Patients With Tuberculosis History
Acronym: INFINITY
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CQAB149BKR01
Record Dates: First submitted 2013-01-25; First posted 2013-01-29 (Estimated); Results first posted 2015-09-18 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Patients With Moderate-to-severe COPD With Destroyed Lung by Tuberculosis
MeSH Terms: interventions — indacaterol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Indacaterol (Experimental): Indacaterol 150 µg once daily
  Interventions: Drug: Indacaterol
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Drug: Control

INTERVENTIONS:
Drug: Indacaterol — Indacaterol 150µg once daily oral inhalation
  Arms: Indacaterol
Drug: Control — Placebo once daily oral inhalation
  Other Names: Placebo
  Arms: Placebo

SUMMARY:
This clinical study will assess efficacy and safety of indacaterol (150㎍ o.d.) in patients with Chronic Obstructive Pulmonary Disease (COPD) with destroyed lung by tuberculosis.

DETAILED DESCRIPTION:
There are few clinical studies in patients with COPD with destroyed lung by tuberculosis because tuberculosis patients are usually excluded from (phase II or III) clinical trials for drug registration although they are not prohibited from prescription of COPD drugs.

This clinical study will assess efficacy and safety of indacaterol (150㎍ o.d.) in patients with COPD with destroyed lung by tuberculosis.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adults aged ≥ 19 years in international age
* Patients with a diagnosis of moderate-to-severe COPD as classified by the GOLD guidelines (2009)
* Patients with at least one finding of destructed pulmonary parenchyma in the chest X-ray and the sum of all legion volumes equivalent to over 1/3 of one lung
* Patients with a history of tuberculosis and no change in the chest imaging test over the past one year
* Patients who can voluntarily sign an Informed Consent Form prior to initiation of any study-related procedure

Exclusion Criteria:

* Pregnant or nursing (lactating) women
* Women of childbearing potential not willing to use effective contraception. However, those who have a negative pregnancy test and agree to use effective contraception can participate. Effective contraception does not include periodical abstinence (e.g. basal body temperature, menstrual cycle contraceptive method, etc) but means use of contraception which must include one of barrier contraceptive methods.

  e.g.) condom (barrier contraceptive method), diaphragms (barrier contraceptive method), oral contraceptives, intrauterine device, Depo injection, etc.
* Patients who have been admitted to hospital for COPD worsening within 6 weeks prior to visit 1
* Patients with a history of respiratory infection within 6 weeks prior to visit 1
* Patients requiring long-term oxygen therapy (>15 hours/1 day) for chronic hypoxemia (it is allowed to use up to a total of 10 out of 24 hours on a PRN basis)
* Patients with a history of asthma
* Unstable ischaemic heart disease, arrhythmia (except for stable ventricular fibrillation) and uncontrolled hypertension
* Patients with a history of long QT syndrome or whose QTc interval measured at Visit 2 is prolonged: >450 ms (males) or >470 ms (females)
* Uncontrolled hypothyroidism and hyperthyroidism
* Hypokalemia: plasma potassium level < 3.0 mEq/L
* Patients with creatinine level ≥2 the upper limit of normal
* Patients with AST/ALT level ≥2 the upper limit of normal
* Patients with lung cancer or a history of lung cancer
* Patients with active cancer or a history of cancer with less than 5 years disease-free survival (whether or not there is evidence of local recurrence or metastases; localized basal cell carcinoma of the skin without metastases is acceptable).
* Patients with a history of hypersensitivity to any of the study drugs or to drugs with similar chemical structures including untoward reactions to sympathomimetic amines or inhaled medication or any component thereof.
* Patients who have had live attenuated vaccinations within 30 days prior to Visit 1
* Patients who have had treatment with investigational drugs, within 30 days or 5 half-lives prior to Visit 1, whichever is longer.
* Patients unable to successfully use a dry powder inhaler device, metered dose inhaler or perform spirometry measurements
* Other cases which are considered ineligible for this clinical study by the principal investigator and subinvestigator

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chul-Gyu Yoo, MD PhD, Principal Investigator — Seoul National University Hospital
Locations (8):
- South Korea (8):
  - Novartis Investigative Site, Anyang-si, Gyeonggi-do
  - Novartis Investigative Site, Koyang-si, Gyeonggi-do
  - Novartis Investigative Site, Jeonju, Jeollabuk-do
  - Novartis Investigative Site, Seoul, Korea
  - Novartis Investigative Site, Koyang, Kyunggi
  - Novartis Investigative Site, Seoul, Seoul
  - Novartis Investigative Site, Incheon
  - Novartis Investigative Site, Seoul

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indacaterol | Placebo
Started | 68 | 68
Safety Set | 68 | 68
Intent to Treat (ITT) | 68 | 67 (One failed to perform primary efficacy evaluation and was excluded, 135 were included in the ITT set)
Completed | 62 | 57
Not Completed | 6 | 11
Not completed — Adverse Event | 1 | 3
Not completed — Consent Withdrawal | 1 | 5
Not completed — major protocol deviation | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Indacaterol | Placebo | Total
Number analyzed (Participants) | 68 | 68 | 136
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.96 (10.90) | 64.62 (9.20) | 64.29 (10.06)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 28 | 51
  Male | 45 | 40 | 85

OUTCOME MEASURES:

1. Primary Outcome: Trough Forced Expiratory Volume in One Second Change
Description: Spirometry was conducted according to internationally accepted standards. Trough FEV1 was defined as the average of the 23 hour 10 minute and 23 hour 45 minute post-dose FEV1 readings. Mixed model used baseline FEV1, FEV1 prior to and 10-15 minutes post inhalation of albuterol, and FEV1 prior to and 1 hour post inhalation of ipratropium as covariate
Time Frame: 8 week
Population: ITT (intent to treat) population included data obtained from all the subjects who were enrolled in the study and received at least one dose of the investigational drug and had primary efficacy endpoint after administration of the investigational drug.
Measure: Mean (Standard Deviation); unit: Liters
Arm/Group | Indacaterol | Placebo
Number analyzed (Participants) | 68 | 67
Liters | 0.08 (0.16) | -0.06 (0.10)
Statistical Analysis 1: Comparison: Indacaterol vs Placebo; Test type: Superiority or Other; p < 0.0001, ANCOVA

2. Secondary Outcome: St. George Respiratory Questionnaire for COPD (SGRQ-C) Change After 8 Weeks of Treatment
Description: The SGRQ-C contains 14 questions divided into two components. Part 1 produces "Symptoms" scores and Part 2 "Activity" and "Impacts" scores. 14 questions which are divided in three domains: "symptom" (question 1-7), "activity" (question 9, 12) and "impact" (question 8, 10, 11, 13 and 14). The total score is 0 to 100 with a higher score indicating greater impairment of health status. Mixed model used baseline SGRQ, FEV1 prior to and 10-15 minutes post inhalation of salbutamol/albuterol, FEV1 prior to and 1 hour post inhalation of ipratropium, and inhaled corticosteroid use at baseline as covariates.
Time Frame: 8 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Indacaterol | Placebo
Number analyzed (Participants) | 68 | 66
Score on a scale | -2.69 (13.00) | -0.33 (16.30)

3. Secondary Outcome: Change From Baseline in Transition Dyspnea Index (TDI) After 8 Weeks of Treatment
Description: TDI focal score is based on three domains: functional impairment, magnitude of task and magnitude of effort. Each domain is scored from -3 (major deterioration) to 3 (major improvement) to give an overall TDI focal score of -9 to 9 with a negative score indicating a deterioration from baseline. A 1 unit difference in the TDI focal score is clinically significant. Mixed model used baseline dyspnoea index, FEV1 prior to and 10-15 minutes post inhalation of albuterol, and FEV1 prior to 1 hour post inhalation of ipratropium as covariates.
Time Frame: 8 week
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Indacaterol | Placebo
Number analyzed (Participants) | 68 | 66
Score on a scale | 1.01 (2.15) | 0.23 (2.38)

4. Secondary Outcome: Incidence of COPD Exacerbation
Description: Number of COPD exacerbation during 8-week treatment. COPD exacerbations are defined as a new onset or worsening of at least one respiratory symptom (i.e. dyspnea, cough, sputum purulence or volume, or wheeze) present for at least 3 consecutive days, documented change or increase in COPD-related treatment due to worsening symptoms or documented COPD-related hospitalizations or emergency room visits.
Time Frame: 8 week
Population: as for outcome 1
Measure: Number; unit: Participants
Arm/Group | Indacaterol | Placebo
Number analyzed (Participants) | 68 | 67
Participants | 3 | 5

ADVERSE EVENTS:
Groups:
- Indacaterol: Indacaterol
- Placebo: Placebo
Arm/Group | Indacaterol | Placebo
Serious Adverse Events (participants affected / at risk) | 3/68 | 1/68
Other Adverse Events (participants affected / at risk) | 9/68 | 13/68
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=68) | Placebo (N=68)
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Indacaterol (N=68) | Placebo (N=68)
Nasopharyngitis (Infections and infestations) | 3 | 4
Upper respiratory tract infection (Infections and infestations) | 3 | 7
COPD Exacerbation (Respiratory, thoracic and mediastinal disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial or disclosure of trial results in their entirety